CLINICAL TRIAL: NCT06451406
Title: Hyaluronic Acid Injection in the Glans Penis Versus Selective Serotonin Reuptake Inhibitors for Lifelong Premature: A Randomized Controlled Trial
Brief Title: Hyaluronic Acid Injection in the Glans Penis Versus Selective Serotonin Reuptake Inhibitors for Lifelong Premature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Waheed Fawzy Abdelrasol, Lecturer of Urology, Faculty of medicine, New Vally University, New Vally, Egypt, New Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240130002
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Selective Serotonin Reuptake Inhibitor; Hyaluronic Acid; Glans Penis; Lifelong Premature
MeSH Terms: interventions — Selective Serotonin Reuptake Inhibitors; Hyaluronic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective serotonin re-uptake inhibitor (Active Comparator): Patients received selective serotonin re-uptake inhibitor (SSRI) as medical treatment for treatment of premature ejaculate.
  Interventions: Drug: Selective serotonin re-uptake inhibitor
- Hyaluronic acid (Experimental): Patients received hyaluronic acid gel injection in the glans penis.
  Interventions: Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Selective serotonin re-uptake inhibitor — Patients received selective serotonin re-uptake inhibitor as medical treatment for treatment of premature ejaculate.
  Arms: Selective serotonin re-uptake inhibitor
Drug: Hyaluronic acid — Patients received injection of glans penis with hyaluronic acid
  Arms: Hyaluronic acid

SUMMARY:
The aim of this study was to compare the effectiveness and safety of selective serotonin reuptake inhibitors (dapoxetine) and hyaluronic acid gel injection in the glans penis for lifelong premature.

DETAILED DESCRIPTION:
Over the past 30 years, the common knowledge of Premature ejaculation (PE) has advanced strikingly. PE is a very common and upsetting sexual male dysfunction. It is disturbing for both partners affecting their sexual experience, reducing their quality of life up to sexual abstinence, causing lack of self-confidence and even depression. It has a prevalence of a variable range, yet it is thought that one third of all males might complain of PE at a certain point throughout their lives and the incidence is rising.

Many treatment modalities have been currently used for PE varying from behavioral therapy to medical treatment and finally surgical therapy. Methods of behavioral therapy are: Squeeze technique and Start/stop technique. Pharmacological therapies include: nonselective and selective SSRIs, topical therapy with anesthetics, PDE5 inhibitors, opioid agonists and others. As for surgical modalities for PE there are several techniques including: glans augmentation, frenectomy, dorsal selective neurectomy, pulsed radiofrequency neuromodulation, removal of foreskin remnants and varicocelectomy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Males.
* Suffering from lifelong premature ejaculation not responding to the behavioral therapy.

Exclusion Criteria:

* Erectile dysfunction.
* Prostatitis.
* Acquired premature ejaculation.
* Addiction.
* Psychiatric disorders (e.g., schizophrenia, bipolar disorder, and other psychoses).
* Historical use of ejaculatory medication within the previous three months.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males suffering from lifelong premature ejaculation not responding to the behavioral therapy
Enrollment: 60 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Intravaginal ejaculation latency time (IELT) | 6 months following treatment
  Intravaginal ejaculation latency time (IELT) is time from initiating sexual activity to ejaculation and used for diagnosis of Long-term premature ejaculation. It was assessed at the 1st, 3rd, and 6th months following treatment.

SECONDARY OUTCOMES:
International index of erectile function-5 (IIEF-5) | 6 months following treatment
  International index of erectile function-5 (IIEF-5) was used for diagnosis of Long-term premature ejaculation and classified into five categories: no (score 22-25), mild (17-21), mild to moderate (12-16), moderate (8-11), and severe (5-7). It was assessed at the 1st, 3rd, and 6th months following treatment.
Index of premature ejaculation (IPE) | 6 months following treatment
  Index of premature ejaculation (IPE) is a 10 item self-administered questionnaire designed to evaluate sexual satisfaction, control and distress in men with premature ejaculation. It diagnosis premature ejaculation (PE) (≤8), possible PE (9 or 10), and no PE (≥11).It was assessed at the 1st, 3rd, and 6th months following treatment.
Patient satisfaction | 6 months following treatment
  Degree of patient satisfaction was assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).
  Degree of patient satisfaction was assessed at the 1st, 3rd, and 6th months following treatment.
Incidence of side effects | 6 months following treatment
  Side effects such as nausea, dizziness, headache, dry mouth, pain at site of injection, ecchymosis, and bullae formation at site of injection were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- New Valley University, New Valley, New Valley Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.